CLINICAL TRIAL: NCT01219894
Title: Frequency Domain Imaging to Determine Stent Strut Coverage and Duration of Anti-Platelet Treatment After Endeavor Stent Placement
Brief Title: Intravascular Optical Coherence Tomography Imaging - Length of Anti-Platelet Therapy After Drug Eluting Stent Placement
Acronym: FDI-DAPT-ZES
Status: Withdrawn | Type: Observational
Why Stopped: Number of patients to meet individual IDE requirements was not obtained.
Sponsor: Emory University (Other)
Collaborators: Medtronic Vascular (Industry); Light Lab Imaging, Inc. (Industry); Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Aloke V. Finn, Principal Investigator, Emory University
Other Study IDs: IRB00045456
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Disease; Stent; Healing; Anti-platelet therapy
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RUTTS Score <30%: Patients with evidence of complete healing of stent at 3 months
- RUTTS<30%: Group with evidence of incomplete healing of the stent

SUMMARY:
Patients who receive drug-coated stents (as opposed to the less frequently used bare metal stents) are currently recommended aspirin plus a thienopyridine such as Plavix, Effient, or Ticlid for one year. These guidelines apply to all patients with drug-coated stents, regardless of the type of stent they received. The purpose of these medications is to prevent a clot at the stent site when there is poor healing of artery tissues over the stent. A clot is a serious concern because it can suddenly block blood flow to the heart and cause a heart attack. These medications have been proven to be helpful in stent patients, but they do have risks. The common side-effects are related to bleeding which in a few patients can be serious. A patient may be at risk for forming a clot if they must put these medications on hold for a surgical procedure to reduce the risk of bleeding. Plavix and Effient are also expensive for patients who are underinsured or uninsured. There is interest is finding a way to show that a patient's stent has healed properly before 12 months and that they can safely stop these medications early.

This study is looking at a way to determine if patients who receive the Endeavor drug-coated stent and who are prescribed aspirin and Plavix can safely stop Plavix at 3 months instead of 12. Previous studies have shown 99.9% coverage of the body's own tissues on an Endeavor stent after 3 months.

A device called an Optical Coherence Tomography (OCT) catheter will be used in this study to look at how much a stent has healed. It allows imaging inside a heart artery and the ability to see the healing of tissues over the stent.

DETAILED DESCRIPTION:
There is a need to find a personalized approach to prescribing dual anti-platelet therapy after a stent is placed in a coronary artery. Stenting involves inserting and expanding a metal tube-shaped device in a heart artery where a blockage is limiting blood flow to the heart muscle. This device stays in the artery permanently and the body's tissues grow over it over time.

Patients in the study will have Optical Coherence Tomography (OCT) imaging done before stent placement and again 3 months later in a follow-up angiography. Patients with sufficient stent healing at 3 months will stop taking Plavix. Patients who have poor stent healing at 3 months will have to continue Plavix through 12 months. Patients will be called once a month during the first year to see how they are doing and if they are taking their prescribed medicines.

Other diagnostic methods that are used when patients have suspected heart blockages include intravascular ultrasound (a device on a catheter that allows ultrasound imaging inside a vessel), fractional flow reserve (a measurement of blood flow to determine if a blockages is serious enough to need treatment), angiography (injection of dye into the arteries to look for narrowing or blockages). These methods are used to look at the severity of heart blockages once a patient already has signs and symptoms. They are not appropriate devices for seeing if a patient's previous stent has healed properly after a certain period of time.

The long-term effectiveness of stenting procedures to treat symptomatic coronary artery disease is limited by the need to take dual anti-platelet therapy (DAPT) with aspirin and plavix to prevent complications related to clot formation within these devices due to incomplete healing of the stented segment. While anti-platelet pharmacologic therapy can minimize this risk, it is associated with an increased risk of serious bleeding events. Currently all patients receiving drug eluting stents (DES) are advised to take plavix for twelve months although a personalized approach for determining the appropriate duration of anti-platelet therapy on a patient by patient basis would reduce both thrombosis and bleeding, thereby improving the long-term safety of coronary revascularization procedures. Optical coherence tomography (OCT) is a new high resolution imaging modality with the potential to discern stent strut healing at follow-up and thus allow for individual tailoring of anti-platelet regimens. Among the commercially available coated stents used in the U.S., the zotarolimus eluting stents (ZES or Endeavor) has demonstrated superior endothelialization and long term safety data in both preclinical and clinical studies and it is very likely earlier discontinuation of anti-platelet therapy is safe. In this trial, patients undergoing ZES placement for symptomatic CAD will undergo 3 months follow-up OCT imaging to determine stent strut healing. Patients demonstrating complete healing will be withdrawn from plavix (with aspirin continued) while those with evidence of incomplete healing will be continued on DAPT for another 9 months. All patients will be followed clinically for another 9 months and intercurrent adverse events recorded. In the end, this research will establish OCT determined stent healing as a surrogate measure for determining optimal anti-platelet therapy following DES implantation.

ELIGIBILITY:
Inclusion Criteria:

* Any patient requiring percutaneous coronary intervention and meeting criteria (as determined by the performing physician) for Endeavor Drug Eluting Stent Placement

Exclusion Criteria:

* Patients requiring >1 stent per treated lesion
* ST segment elevation MI (STEMI)
* inability to comply with study follow-up including 12 months of DAPT
* current or planned pregnancy (for women of childbearing age)

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing percutaneous transluminal coronary intervention (PTCI) for treatment of de novo native vessel coronary artery disease with a single DES (EndeavorTM, zotarolimus, Medtronic Vascular) will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Ratio of Uncovered to Total Stent Struts Per Cross Section (RUTTS) score of ≤30% of the target stent as determined by OCT pullback of the target stent | 3 months
  Primary Endpoint: The primary endpoint of this trial will be the frequency of near complete healing 3 months after Endeavor placement defined as a Ratio of Uncovered to Total Stent Struts Per Cross Section (RUTTS) score of ≤30%.

SECONDARY OUTCOMES:
death | 1 year
  Occurrence of events after 3-month follow-up in the group with OCT guided early discontinuation of DAPT versus those adhering to standard of care (i.e. 12 months of DAPT). Events will be defined as death, stent thrombosis (Academic Research Consortium definition), myocardial infarction (defined as any evidence of troponin elevation above the upper limit of normal), and bleeding (TIMI Bleeding Classification (table 1)). We will also examine the relationship between underlying plaque morphology and 3 month follow-up OCT determined strut coverage.
Stent Thrombosis | 1 year
  As defined by the Academic Research Consortium definition.
myocardial infarction | 1 year
  Defined as any troponin elevation above the upper limit of normal
Bleeding | 1 year
  As defined by the TIMI Bleeding Classification.

CONTACTS AND LOCATIONS:
Overall Officials: Aloke Finn, MD, Principal Investigator — Emory University

REFERENCES:
- [Background] Finn AV, Joner M, Nakazawa G, Kolodgie F, Newell J, John MC, Gold HK, Virmani R. Pathological correlates of late drug-eluting stent thrombosis: strut coverage as a marker of endothelialization. Circulation. 2007 May 8;115(18):2435-41. doi: 10.1161/CIRCULATIONAHA.107.693739. Epub 2007 Apr 16. PMID 17438147
- [Background] Kim JS, Jang IK, Fan C, Kim TH, Kim JS, Park SM, Choi EY, Lee SH, Ko YG, Choi D, Hong MK, Jang Y. Evaluation in 3 months duration of neointimal coverage after zotarolimus-eluting stent implantation by optical coherence tomography: the ENDEAVOR OCT trial. JACC Cardiovasc Interv. 2009 Dec;2(12):1240-7. doi: 10.1016/j.jcin.2009.10.006. PMID 20129551